CLINICAL TRIAL: NCT04751032
Title: Chinese Nutritional Risk Screening and Intervention Registration Study in Geriatric Patients
Acronym: CNRSIS
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: NCT2020090120210601
Record Dates: First submitted 2021-01-23; First posted 2021-02-11 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2020-10

CONDITIONS: Malnutrition; Old Age
Keywords: malnutrition; older adults; adverse outcomes; nutrition intervention
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-center observational study, led by the Department of Geriatrics, Peking Union Medical College Hospital, with 99 tertiary hospitals as sub-centers. Patients in the geriatrics department from September 2020 to September 2021 are consecutively enrolled .Basic information and nutritional risk assessment is registered and the outcome within 90 days after hospitalization will be recorded.Daily energy, protein and fiber are 75% of the target amount as the standard for feeding.

DETAILED DESCRIPTION:
This study is a multi-center observational study.Patients in the geriatrics department from September 2020 to September 2021 are consecutively enrolled .The patients' basic information, nutritional assessment, diet and blood biochemical indicators after hospitalization will be registered.The status of nutritional treatment and rehabilitation training and whether there is any adverse outcome when discharged from the hospital will be recorded. Daily energy, protein and fiber are 75% of the target amount as the standard for feeding.The diet, exercise status and adverse outcomes of participants within 90 days after hospitalization will be followed up through outpatient, telephone or remote consultation.Primary endpoint-the impact of nutritional therapy (energy, protein, dietary fiber compliance or failure) on mortality, new infections, falls and readmissions in elderly hospitalized patients within 90 days after hospitalization; secondary endpoints-the change of the nutrition indicators, the physical function and quality of life of the participants within 90 days after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 years old in geriatrics;
* Expected hospitalization ≥4 days;
* Patients with NRS 2002≥3 points;
* Sign informed notice.

Exclusion Criteria:

* End-stage patients (estimated survival time ≤ 3 months);
* Transfer to other departments during hospitalization;
* Contraindications to nutritional therapy (such as hemodynamic instability);
* Have participated in other nutritional research projects.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients in the geriatrics/geriatrics department of tertiary hospitals from September 2020 to September 2021 are consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of mortality | within 90 days after hospitalization
  all cause mortality
Number of Participants with respiratory, urinary or gastrointestinal infections diagnosed by clinicians | within 90 days after hospitalization
  Any infection diagnosed by a formal medical institution.Infections that require a doctor's prescription of antibiotics indicated in the medical records or diagnosis reports provided by the participants, including the respiratory tract, urinary tract, gastrointestinal tract, etc.The report or diagnosis certificate has relevant evidence, for example, the test indicates that the white blood cell is increased or the high-sensitivity C-reactive protein is increased.
Number of Participants with unplanned hospitalization for acute illness | within 90 days after hospitalization
  Visits reported by participants because of an acute illness rather than regular visits.Hospital stays longer than 48 hours will be counted, but outpatient visits will not be counted.
Number of Participants with fall | within 90 days after hospitalization
  Any falls reported by the participants within 90 days will be recorded. The cause of the fall and whether it is accompanied by a fracture shall be recorded.

SECONDARY OUTCOMES:
Number of Participants with the albumin changes | Within 90 days after hospitalization
  The albumin level of the 90-day follow-up and baseline will be measured in the unified laboratory using the same monitoring method, and the changes are used as the evaluation index of nutrition
Number of Participants with the physical function changes assessed by katz activity of the daily living（ADL） | Within 90 days after hospitalization
  The Katz scale goes by the basics to evaluate a patient's level of independence or dependence.The 90-day follow-up and baseline ADL scores will be evaluated by trained elderly doctors, and the changes are used as the evaluation indicators for functional changes
Number of Participants with the quality of the life changes according to the EuroQol Five Dimensions Questionnaire（EQ-5D） | Within 90 days after hospitalization
  the change of the score of the EQ-5D assessed by the participants.EQ-5D, EuroQol Five Dimensions Questionnaire, is a set of standardized scales for measuring health status. EQ-5D was developed by the European Society for Quality of Life (EuroQol), which can provide a simple and universal health measurement method. In the description part, five dimensions will be used to describe the health status. The five dimensions are: Mobility, Self-care, Usual Activities, Pain/Discomfort ), Anxiety/Depression. The questionnaire requires respondents to choose the most suitable option in each dimension according to their health status.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Liu, MD &PHD, Principal Investigator — Department of Geriatrics,Peking Union Medical College Hospital
Locations (1):
- Department of Geriatrics,Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li M, Jiang S, Li J, Chen X, Ma L, Guo Q, Wang Y, Luo L, An L, Wu Y, Huang W, Yuan L, Wang L, Ding X, Zhao X, Zhang Z, Zhang H, Wu Y, Yang R, Liu Y, Cao J, Liu X. Effectiveness and safety of oral nutrition in older patients with moderate dysphagia: a real-world cohort study in geriatric inpatients. BMC Geriatr. 2025 Jul 31;25(1):571. doi: 10.1186/s12877-025-06175-2. PMID 40745263